CLINICAL TRIAL: NCT06617403
Title: Can Pre-operative Characteristics Predict Failure of Supraglottic Airway to Tracheal Tube? A Machine Learning Algorithm (ERICA)
Brief Title: Pre-operative Characteristics for Prediction of Supraglottic Airway Failure Using Machine Learning (ERICA)
Acronym: ERICA
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Ulm (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Flora Scheffenbichler, Dr. med., University Hospital Ulm
Other Study IDs: ERICA
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Anesthesia, General; Postoperative Complications; Laryngeal Masks; Treatment Failure
Keywords: "Neural Networks, Computer Artificial Intelligence"[Mesh]; "Laryngeal Masks"[Mesh]; "Treatment Failure"[Mesh]; "Treatment Outcome"[Mesh]; "Risk Factors"[Mesh]
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non — non

SUMMARY:
Supraglottic airway devices (SGA) are a safe and well-established technique for airway management. Nowadays, up to 60% of general anaesthetics performed in European countries use SGA. In 0.2-4.7% SGA fail and require conversion to tracheal tubes.

The ERICA study will use artificial intelligence methods to develop a model that can predict the risk of an unplanned SGA conversion based on pre-operative characteristics available during the premedication visit.

DETAILED DESCRIPTION:
An intraoperative change of procedure not only leads to time delays but also time delays, but also involves measures that are stressful for the patient, such as deepening the anaesthesia and manipulating the airway again.

Therefore, the objective of ERICA is to develop a machine learning algorithm based on preoperative information 1) that can accurately predict the risk of an unplanned SGA conversion and 2) identifies characteristics leading to conversion from SGA to tracheal tube.

I. Developing the model

• The final dataset will be split in a training, testing, and validation cohort. Five models will be created to predict intraoperative conversion from SGA to tracheal tube including generalized linear models (GLM), deep learning, distributed random forest (DRF), xgboost and gradient boosting machine (GBM). Then, a stacked ensemble model will be constructed through combination of the five models. Finally, the best artificial intelligence model will be chosen.

II. Identify characteristics leading to the airway conversion and categorisation.

* Intraoperative changes of the patient's position can alter the risk of conversion, therefore operations with positional changes should be considered
* Identify patient- and procedure-dependent characteristics that lead to conversion from SGA to tracheal tube and their importance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) receiving general anaesthesia for non-cardiac surgery with a supraglottic airway device

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) receiving non-cardiac surgery using a supraglottic airway device
Sampling Method: Non-Probability Sample
Enrollment: 44000 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of unplanned SGA conversion | intraoperative

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Ulm, Ulm, Baden-Wurttemberg
  - Technical University Munich, Munich, Bavaria